CLINICAL TRIAL: NCT04538222
Title: An Effectiveness Study of Workplace Physical Activity Intervention for Staff in a Hospital Setting
Brief Title: Workplace Physical Activity Intervention
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202007050RIND
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2020-08

CONDITIONS: Health Promotion
Keywords: workplace; health promotion
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physical activity — aerobic exercise, muscle strength and stretching, nutrition education

SUMMARY:
In this study, it investigates the effectiveness of workplace physical activity intervention for staff in a 100-bed hospital in Taipei City, Taiwan. The physical activity program takes group coaching and includes aerobic exercise, muscle strength and stretching in combination with nutrition education. The duration of the program is three months (8 sessions per month). The subjects of the study were recruited from full-time employees working at the hospital who attend the program. The recruited employees can take part in the program freely and chose types of activity by themselves. This study measures body mass index, muscle strength, body fat percentage, muscle strength, body mass index, daily energy expenditure, and exercise self-efficacy as the baseline. After 3-month program, we will evaluate the effectiveness of the program. The result is anticipated the greater frequent attendance, the more obvious effectiveness in outcomes.

DETAILED DESCRIPTION:
A three-month group coaching physical activity program in combination with nutrition education was developed for full-time employees working on a 100-bed hospital in Taipei City, Taiwan. Due to the setting that employees can take part in the program freely and chose types of activity by themselves. So participants may have various intensity of participation. This study aims to evaluate the effectiveness of pre- and post- 3-month workplace physical activity programs in body fat percentage, Muscle strength, body mass index, daily energy expenditure, and exercise self-efficacy. One group pretest-posttest design was used for the study by convenience sampling technique. Subjects were recruited from participants of the program. The intervention consists of : (1)education on nutrition: 2 times per month for 3 months, 1 hour/time ; and (2)physical activity: a three-month group coaching program (24 sessions), including three types of exercise courses such as aerobic exercise, muscle strength and stretching. All analyses were performed using Statistics Analysis System version 9.3 and the effects of the intervention were assessed by the paired t-test. Multiple regression analysis was used to determine the contribution of attendances of activities and behavior change stage to effectiveness of workplace physical activity. The level of significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* full-time employees
* Complete the informed consent

Exclusion Criteria:

* With pacemaker
* accepted or are participating participate other weight control related research or interventional medicine

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals who participate hospital self-developed workplace physical activity
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Body fat percentage at 3 months | baseline, 3 month after intervention
  Body fat percentage was the total mass of fat divided by total body mass, multiplied by 100. Estimate for body fat percentage was measured by dual frequency bio-electric impedance(BIA) body composition analyzer.
Change from Baseline Muscle strength at 3 months | baseline, 3 month after intervention
  Muscle strength was assessed by hand grip strength using a grip strength dynamometer. The grip strength dynamometer can measure range from 5 to 100 kg. During the measurement, the subject stood upright and was asked to hold the grip with the dynamometer with the greatest strength. Take the maximum value after two measurements.
Change from Baseline exercise self-efficacy at 3 months | baseline, 3 month after intervention
  The five-item self-efficacy questionnaire designed to measure confidence in one's ability to persist with exercising in various situations which included the following: tired, bad mood, don't have the time, on vacation, raining or snowing. An 7-point scale was used to rate each item of self-efficacy, scores range from 5 "not at all confident" to 35 "very confident". A score of 0 means "extremely low self-efficacy" and a score of 35 means" "extremely high self efficacy"
Change from Baseline exercise behavior change stage at 3 months | baseline, 3 month after intervention
  exercise behavior change stage

SECONDARY OUTCOMES:
Change from Baseline body mass index at 3 months | baseline, 3 month after intervention
  Body mass index (BMI) was calculated as body weight (kg) divided by the square of the body height (meter) (m2). BMI was assessed using a body composition analyzer.
Change from Baseline Daily energy expenditure at 3 months | baseline, 3 month after intervention
  Daily energy expenditure as an estimate of total kilo-calories of energy expended per day. Calculation from the seven-day physical activity recall questionnaire. Subjects were asked to list total activities in each category and quantifying the time spent (hour) in each activity over a seven-day period. Activities were classified by their energy requirements, expressed in terms of Metabolic Equivalent of Task (MET). Sleep = 1 MET; light activity = 1.0-2.9 MET (MET level: 1.5); moderate activity = 3.0-5.0 MET (MET level: 4); hard activity =5.1-6.9 MET (MET level: 6); very hard activity = 7.0 or greater MET (MET level: 10). Each activity's total kilo-calories of energy expended per day was calculated by the following equation: activity MET * times of having activity time(hours)*body weight(kg)/7 (day).

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Taipei, 新店區